CLINICAL TRIAL: NCT00729664
Title: A Phase 1, Multidose Study of BMS-936559 (MDX-1105) Administered Every 14 Days in Subjects With Selected Advanced or Recurrent Solid Tumors
Brief Title: Multiple Ascending Dose (MDX1105-01)
Acronym: Anti-PDL1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA210-001; MDX1105-01 (Other: BMS)
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Cancer, Multiple Indications
MeSH Terms: conditions — Neoplasms | interventions — BMS-936559

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Anti-PDL-1 antibody (Arm 1) (Experimental): BMS-936559 (MDX-1105)
  Interventions: Biological: Anti-PDL-1 antibody
- Anti-PDL-1 antibody (Arm 2) (Experimental): BMS-936559 (MDX-1105)
  Interventions: Biological: Anti-PDL-1 antibody
- Anti-PDL-1 antibody (Arm 3) (Experimental): BMS-936559 (MDX-1105)
  Interventions: Biological: Anti-PDL-1 antibody
- Anti-PDL-1 antibody (Arm 4) (Experimental): BMS-936559 (MDX-1105)
  Interventions: Biological: Anti-PDL-1 antibody
- Anti-PDL-1 antibody (Arm 5) (Experimental): BMS-936559 (MDX-1105)
  Interventions: Biological: Anti-PDL-1 antibody

INTERVENTIONS:
Biological: Anti-PDL-1 antibody — Solution, Intravenous, 0.1 mg/kg, Every 14 days, 3 doses per each cycle of 42 days, 16 cycles/48 doses depending on response
  Other Names: BMS-936559; MDX 1105
  Arms: Anti-PDL-1 antibody (Arm 1)
Biological: Anti-PDL-1 antibody — Solution, Intravenous, 0.3 mg/kg, Every 14 days, 3 doses per each cycle of 42 days, 16 cycles/48 doses depending on response
  Other Names: BMS-936559; MDX 1105
  Arms: Anti-PDL-1 antibody (Arm 2)
Biological: Anti-PDL-1 antibody — Solution, Intravenous, 1 mg/kg, Every 14 days, 3 doses per each cycle of 42 days, 16 cycles/48 doses depending on response
  Other Names: BMS-936559; MDX 1105
  Arms: Anti-PDL-1 antibody (Arm 3)
Biological: Anti-PDL-1 antibody — Solution, Intravenous, 3 mg/kg, Every 14 days, 3 doses per each cycle of 42 days, 16 cycles/48 doses depending on response
  Other Names: BMS-936559; MDX 1105
  Arms: Anti-PDL-1 antibody (Arm 4)
Biological: Anti-PDL-1 antibody — Solution, Intravenous, 10 mg/kg, Every 14 days, 3 doses per each cycle of 42 days, 16 cycles/48 doses depending on response
  Other Names: BMS-936559; MDX 1105
  Arms: Anti-PDL-1 antibody (Arm 5)

SUMMARY:
Collection of survival data, evaluation of PDL-1 expression in tumors, and evaluation of PD-L1 receptor occupancy in peripheral blood has been added.

DETAILED DESCRIPTION:
This is an open label, multicenter, dose escalation and multidose study of MDX-11-5, a fully human monoclonal IgG4 antibody targeting the Programed Death-Ligand 1 (PD-L1).

The study will consist of 3 periods: Screening (up to 28 days), Treatment (up to 16 six-week cycles), and Follow-up (up to 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1
* The malignancies include relapsed/refractory renal cell carcinoma, non-small cell lung cancer, colorectal adenocarcinoma, malignant melanoma, advanced/metastatic epithelial ovarian cancer, gastric cancer, pancreatic cancer and breastcancer
* Must have measurable disease

Exclusion Criteria:

* Prior therapy with an anti-PD 1, anti-PDL 1, or anti-Cytotoxic T-Lymphocyte Antigen 4 antibody (or any other agents that target T-cell co-stimulation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2009-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety, maximum tolerated dose (MTD) and dose-limiting toxicity(DLT)of MDX-1105 | Weekly
Safety, maximum tolerated dose (MTD) and dose-limiting toxicity(DLT)of MDX-1105 | Bi-weekly

SECONDARY OUTCOMES:
Preliminary efficacy in solid tumors on the basis of objective responses | Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (11):
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - University Of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - University Of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oncology Consultants, Pa, Houston, Texas
  - The University Of Texas, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

REFERENCES:
- [Derived] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx